CLINICAL TRIAL: NCT06829186
Title: Effect of Curcumin on the Reduction of Cellular Inflammation Markers in Hemodialysis Patients
Brief Title: The Effect of Curcumin on Inflammatory Markers in Hemodialysis Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Mariana Chávez-Tostado, Doctor in Multidisciplinary Health Research, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: curcumin_hemodialysis; CEI 100/25 (Registry Identifier: CUR/HEMOD-FAA)
Record Dates: First submitted 2025-01-27; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis
Keywords: CURCUMIN; Hemodialysis; INFLAMMATION
MeSH Terms: conditions — Inflammation | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- case group (Experimental): curcumin capsules 500 mg every 8 hours for 12 weeks
  Interventions: Dietary Supplement: Curcumin (Longvida™)
- control group (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin (Longvida™) — patients will be suplemented during 3 months with longvida, 2 cap /8 hours
  Arms: case group
Drug: Placebo — one capsules every 8 hours during 12 weeks
  Arms: control group

SUMMARY:
The goal of this clinical trial is to learn if curcumin can lower the inflammation in participants with chronic kidney disease (CKD) undergoing hemodialysis (HD).

The main questions it aims to answer are:

Does curcumin lower can lower profinflamatory markers in participants with CKD on HD?

Researchers will compare curcumin to a placebo (a look-alike substance that contains no drug) to see if curcumin works to help the treatment in participants with CKD on HD.

Researchers will compare nutritional status and side effects after taking the supplement.

Participants will:

Take the curcumin or a placebo twice a day for 3 months Visit the clinic once every week for checkups and tests.

DETAILED DESCRIPTION:
1. Study Title:

   "Effect of Curcumin on the Reduction of Cellular Inflammation Markers in Hemodialysis Patients"
2. Study Design:

   Type: Randomized, double-blind, placebo-controlled clinical trial.
   * Setting: Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde," Mexico.
   * Participants: 34 CKD patients on hemodialysis or peritoneal dialysis, aged 18+.
   * Intervention: Patients will receive either curcumin (500 mg capsules, 3 times daily) or placebo for 12 weeks with pre- and post-intervention assessments.
3. Objectives:

   Primary Objective: To evaluate the effect of curcumin supplementation on inflammatory markers (TNF-α, IL-1β, IL-6, and CRP) in hemodialysis patients.

   Secondary Objectives:
   * To assess changes in renal metabolites (creatinine, urea, proteinuria).
   * To monitor nutritional status (weight, BMI, muscle mass, dynamometry).
   * To identify potential side effects or adverse reactions associated with curcumin supplementation.
4. Study Population:

   Inclusion Criteria:
   * Patients aged 18 years or older.
   * Clinically stable and receiving hemodialysis for at least 3 months prior to enrollment.
   * Willing to provide informed consent.

   Exclusion Criteria:
   * Active malignancy, severe infections, or systemic inflammatory diseases.
   * Liver disease (ALT/AST > 3x upper limit of normal).
   * Use of immunosuppressants, corticosteroids, or experimental drugs within the last month.
   * Pregnancy, smoking, or allergies to curcumin.
   * Recent antibiotic use (within the last 3 months).
5. Sample Size:

   Calculation: Based on a previous study (Afshar et al., 2020), a sample size of 17 patients per group (34 total) was determined to detect a significant difference in CRP levels with 80% power and a 20% dropout rate.
6. Randomization and Blinding:

   Randomization: Patients will be randomly assigned to either the curcumin or placebo group using sealed, opaque envelopes.

   Blinding: Both participants and investigators will be blinded to the treatment allocation. The placebo capsules will be identical in appearance to the curcumin capsules.
7. Intervention:

   * Curcumin Group: Patients will receive 500 mg curcumin capsules (Longvida® with 20% curcuminoids) two times daily (total of 1 g/day) for 12 weeks.
   * Placebo Group: Patients will receive identical-looking placebo capsules (containing starch) on the same schedule.

   Adherence Monitoring: Patients will be provided with a calendar to track capsule consumption. Adherence will be considered good if ≥80% of capsules are consumed.
8. Data Collection:

   * Baseline and Post-Intervention Assessments:
   * Inflammatory Markers: TNF-α, IL-1β, IL-6, and CRP levels will be measured using ELISA.
   * Renal Function: Serum creatinine, urea, proteinuria, and other renal markers will be assessed.
   * Nutritional Status: Weight, height, BMI, body composition (fat and muscle mass), and handgrip strength (dynamometry) will be measured.
   * Dietary Habits: A 3-day dietary diary will be used to assess protein, fat, fiber, sodium, potassium, and phosphorus intake.
   * Adverse Events: Any side effects or adverse reactions will be recorded during weekly follow-ups.
9. Laboratory Procedures:

   * Blood Samples: Collected before and after the intervention. Samples will be centrifuged and stored at -80°C for biomarker analysis.
   * ELISA Analysis: Inflammatory markers (TNF-α, IL-1β, IL-6, CRP) will be quantified using commercially available ELISA kits.
   * Renal Function Tests: Performed in the hospital's clinical laboratory using standard methods.
10. Statistical Analysis:

    -Descriptive Statistics: Mean, median, standard deviation, and frequencies will -be calculated for continuous and categorical variables.

    Inferential Statistics:
    * Normality will be assessed using Kolmogorov-Smirnov or Shapiro-Wilk tests.
    * Parametric tests (t-tests) or non-parametric tests (Mann-Whitney U) will be used to compare groups.
    * Chi-square or Fisher's exact tests will be used for categorical variables.
    * Changes in inflammatory markers and renal function will be analyzed using paired tests (pre- vs. post-intervention).

    Software: SPSS (version 17.0) and GraphPad Prism (version 10.3.0) will be used for data analysis.
11. Ethical Considerations:

    * Approval: The study protocol has been approved by the Ethics Committee of the Antiguo Hospital Civil de Guadalajara.
    * Informed Consent: All participants will provide written informed consent before enrollment.
    * Confidentiality: Patient data will be anonymized and stored securely. Only the research team will have access to identifiable information.
    * Participant Rights: Participation is voluntary, and patients may withdraw at any time without affecting their medical care.
12. Timeline:

    * May-Oct 2024: Literature review and protocol development.
    * Jan-Mar 2025: Ethical approval and patient recruitment.
    * Mar-Dec 2026: Intervention period and data collection.
    * Dec 2026: Data analysis and manuscript preparation.
    * 2027: Publication and dissemination of results.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes undergoing dialysis or hemodialysis.
* Aged 18 years or older.
* Clinically stable and receiving hemodialysis or dialysis for at least three months before study enrollment.
* Continuation of pharmacotherapy as prescribed by their physician.
* Regular use of antioxidant supplements and turmeric consumption.
* Signed written informed consent.

Exclusion Criteria:

* Active malignant disease (diagnosed within the past five years).
* Critical illness requiring respiratory or circulatory support.
* Severe congestive heart failure (NYHA class IV).
* Severe chronic systemic infectious or inflammatory disease.
* Severe liver disease.
* Known allergy to study products.
* Treatment with immunosuppressants or experimental drugs in the past month.
* Use of anti-inflammatory corticosteroids.
* Scheduled kidney transplant during the study.
* Pregnant patients.
* Active smokers.
* Autoimmune diseases, cancer, severe infections, or AIDS.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Interleukin Interleukin-6 | before supplementation
  basal meassurement of Interleukin-6 in nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)
Interleukin Interleukin-6 | after 3 months of supplementation
  final meassurement of Interleukin-6 nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)
TNF-α: Tumor Necrosis Factor-alpha | before supplementation
  basal meassurement of TNF-α in nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)
TNF-α: Tumor Necrosis Factor-alpha | after 3 months of supplementation
  final meassurement of TNF-α in nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)
IL-1β: Interleukin-1 beta | before supplementation
  basal meassurement of IL-1β in nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)
IL-1β: Interleukin-1 beta | after 3 months of supplementation
  final meassurement of IL-1β in nanometers using the Enzyme-Linked Immunosorbent Assay (ELISA)

SECONDARY OUTCOMES:
Urea | before supplementation
  Urea meassurement in mg/dL using a biochemistry analyzer
Urea | after 3 months of supplementation
  Urea meassurement in mg/dL using a biochemistry analyzer
leukocyte count | before supplementation
  leukocyte count (cells/µL) using an automated blood cell counter
leukocyte count | after 3 months of supplementation
  leukocyte count (cells/µL) using an automated blood cell counter
neutrophil/lymphocyte ratio (NLR) | before supplementation
  NLR (neutrophil/lymphocyte count) using a hematology analyzer.
neutrophil/lymphocyte ratio (NLR) | after 3 months of supplementation
  NLR (neutrophil/lymphocyte count) using a hematology analyzer.
lymphocyte/platelet ratio (LPR) | before supplementation
  LPR (lymphocyte/platelet count) using a hematology analyzer.
lymphocyte/platelet ratio (LPR) | after 3 months of supplementation
  LPR (lymphocyte/platelet count) using a hematology analyzer.
erythrocyte sedimentation rate (ESR) | before supplementation
  ESR (mm/h) using a Westergren ESR analyzer
erythrocyte sedimentation rate (ESR) | after 3 months of supplementation
  ESR (mm/h) using a Westergren ESR analyzer
serum albumin | before supplementation
  serum albumin in g/dL using a biochemistry analyzer
serum albumin | after 3 months of supplementation
  serum albumin in g/dL using a biochemistry analyzer
Weight | before supplementation
  Weight of partipants (kg) using a tanita BC 601® scale
Weight | after 3 months of supplementation
  Weight of partipants (kg) using a tanita BC 601® scale
body mass index (BMI) | before supplementation
  BMI of patients (weight/height*height)
BMI | after 3 months of supplementation
  BMI of patients (weight/height*height)
body fat percentage | before supplementation
  body fat percentage of patients (%) using a tanita BC 601® scale
body fat percentage | after supplementation
  body fat percentage of patients (%) using a tanita BC 601® scale
muscle mass | before supplementation
  muscle mass of patients (kg) using a tanita BC 601® scale
muscle mass | after 3 months of supplementation
  muscle mass of patients (kg) using a tanita BC 601® scale
hand grip strenght | before supplementation
  hand grip strenght of patients using a dynamometer (kg), (Jamar Plus Digital Hand Dynamometer)
hand grip strenght | after 3 months of supplementation
  hand grip strenght of patients using a dynamometer (kg), (Jamar Plus Digital Hand Dynamometer)

IPD SHARING:
Plan to Share IPD: No
results will be used for future studies

REFERENCES:
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Cozzolino M, Galassi A, Pivari F, Ciceri P, Conte F. The Cardiovascular Burden in End-Stage Renal Disease. Contrib Nephrol. 2017;191:44-57. doi: 10.1159/000479250. Epub 2017 Sep 14. PMID 28910790